CLINICAL TRIAL: NCT02951325
Title: Prospective Randomized Trial of Adjuvant Radiotherapy Following Surgery and Chemotherapy in Muscle Invasive Transitional Cell Carcinoma of Urinary Bladder
Brief Title: Bladder Cancer Adjuvant Radiotherapy Trial
Acronym: BART
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Vedang Murthy, Professor and Radiation Oncologist, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BART
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Bladder Cancer; Urothelial Carcinoma Bladder
Keywords: adjuvant RT
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard (No Intervention): Surgery +/- chemotherapy only
  * Surgery (Standard/routine care) Cysto-prostatectomy and pelvic nodal dissection as part of their standard care.
  * Chemotherapy All patients following cysto-prostatectomy (inclusive of those received neo-adjuvant chemotherapy) will receive upto 4 cycles of adjuvant chemotherapy if medically fit for the same. The chemotherapy regimen, doses and schedule will be as per standard institutional practice. No concomitant chemotherapy with radiotherapy is recommended.
  No radiation therapy will be given.
- Test (Experimental): Surgery +/- chemotherapy as per standard arm and Radiation therapy as experimental intervention
  Radiation Therapy:
  All patients will be treated with conformal radiotherapy technique with intensity modulated radiotherapy with or without image guidance. The radiotherapy will start within 8 weeks from the date of surgery if adjuvant chemotherapy has not been planned. The radiotherapy will start within 4 weeks from the date of last chemo cycle, in patients who will be given adjuvant chemotherapy.
  Dose Prescription:
  •50.4 Gray (Gy) in 28 fractions (1.8Gy/#) will be prescribed for the nodal PTV. In case of R1 and/or R2 resection dose to the pelvic nodes and tumour bed may be increased to 54-56 Gy in 28 fractions depending on the constraints achieved during planning.
  Patient assessments: Clinical assessment for toxicity evaluation and disease status. QOL evaluation of the patients.
  Interventions: Other: Adjuvant RT

INTERVENTIONS:
Other: Adjuvant RT — Radiation therapy:
  All patients will be offered conformal technique with IMRT +/- image guidance. The adjuvant RT will start within 8 weeks from the date of surgery if chemotherapy not planned or 4 weeks from the date of last adjuvant chemo cycle.
  Dose:
  •50.4 Gray (Gy) in 28 fractions (1.8Gy/#) for the nodal PTV. For R1 and/or R2 resection increased to 54-56 Gy in 28 fractions based on the constraints achieved during planning.
  Patient assessments:
  Clinical:
  * Toxicity:
    1. Weekly RT with toxicity scoring.
    2. RTOG toxicity criteria at baseline, 6-8 weeks post RT and f/b 3 monthly x 2 years and 6 monthly x 5 years.
    3. QOL will be assessed at baseline f/b 3-6 monthly.
  * Disease evaluation:
    i. first f/u all patients will be at 6-8 week to assess toxicity. ii. Clinical evaluation of the disease will be done at each f/u visit. iii. CT scan (abdomen and pelvis) 6 monthly from visit 2 onwards up to 2 years f/b 12 monthly or as clinically indicated.
  Arms: Test

SUMMARY:
Aim and objectives:

This trial aims to evaluate the role of adjuvant radiotherapy following chemotherapy in patients with high-risk features on histo-pathology after radical surgery for transitional cell carcinoma of urinary bladder

DETAILED DESCRIPTION:
Treatment details:

Surgery(Standard/routine care) All patients would have undergone radical surgery in the form of a cysto-prostatectomy and pelvic nodal dissection as part of their standard care. Patients would also have a urinary diversion (Ileostomy) or a continent neo bladder.

Chemotherapy All patients following cysto-prostatectomy will receive upto 4 cycles of adjuvant chemotherapy if medically fit for the same. Those patients who received neoadjuvant chemotherapy, will receive additional chemotherapy cycle after surgery to a total of 4 cycles if found suitable. The chemotherapy regimen, doses and schedule will be as per standard institutional practice using Platinum based chemotherapy. No concomitant chemotherapy with radiotherapy is recommended.

Radiation therapy:

All patients will be treated with conformal radiotherapy technique with intensity modulated radiotherapy with or without image guidance. The radiotherapy will start within maximum of 8 weeks from the date of surgery if adjuvant chemotherapy has not been planned. If adjuvant chemo planned the patients will receive radiotherapy within 4 weeks of the last chemo cycle.

Dose Prescription:

50.4Gray (Gy) in 28fractions (1.8Gy/#) will be prescribed for the nodal PTV. In case of R1 and/or R2 resection dose to the pelvic nodes and tumour bed may be increased to 54-56Gy in 28 fractions depending on the constraints achieved during planning.

Clinical assessment:

1. Toxicity will be assessed by

   1. Weekly physician assessment during RT with scoring of toxicity.
   2. RTOG toxicity criteria at baseline, 6-8 weeks post RT and at 3 monthly thereafter for 2 years and 6 monthly thereafter for 5 years.
   3. QOL will be assessed at baseline and 3-6 monthly thereafter
2. Disease evaluation The first follow up all patients will be done at 6-8 week to assess toxicity. Clinical evaluation of the disease will be done at each follow up visits by clinical examination. CT scan of the abdomen and pelvis will be done 6 monthly from second visit onwards up to 2 years and 12 monthly thereafter or whenever clinically indicated as decided by the physician.

ELIGIBILITY:
Inclusion Criteria:

All patients should have undergone radical cystoprostatectomy for bladder cancer Patients with any of the below high risk features on histolopathology

* Lymph Node positive with or without perinodal extension (PNE)
* Cut-margin positive,
* pT3 and pT4 disease,
* Number of nodes dissected at surgery < 10 All patients irrespective of the final pathology if they have received neo-adjuvant chemotherapy prior to surgery for any of the following T3 T4 stage N1-3 stage No evidence of distant metastasis including para-aortic nodal metastasis KPS ≥ 70 Signed study specific consent form Adequate hepatic, renal and hematologic parameters

Exclusion Criteria:

* Contraindication to pelvic radiotherapy like inflammatory bowel disease
* Uncontrolled diabetes or hypertension
* Uncontrolled cardiac or respiratory co morbidity
* Prior history of therapeutic irradiation to pelvis
* Patient unwilling and unreliable for follow up and QoL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2016-06-02 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2030-04-13 (Estimated)

PRIMARY OUTCOMES:
Improvement in loco-regional relapse free survival (LRFS) | 2 year

SECONDARY OUTCOMES:
Disease free survival (DFS) | two and five years
Overall survival(OS) | two and five years
RT toxicity (acute and late) | 6 months and 2 years
  RT toxicity will be measured using RTOG and CTCAE grading scale
QOL | 2 years
  FACT questionnaire will be used to assess QOL.
Patterns of failure | 2 years
  The local, regional and distant metastasis rates will be assessed with 6 monthly CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Murthy V, Maitre P, Singh M, Pal M, Arora A, Pujari L, Kapoor A, Pandey H, Sharma R, Gudipudi D, Joshi A, Prabhash K, Noronha V, Menon S, Mehta P, Bakshi G, Prakash G. Study Protocol of the Bladder Adjuvant RadioTherapy (BART) Trial: A Randomised Phase III Trial of Adjuvant Radiotherapy Following Cystectomy in Bladder Cancer. Clin Oncol (R Coll Radiol). 2023 Sep;35(9):e506-e515. doi: 10.1016/j.clon.2023.04.010. Epub 2023 May 5. PMID 37208232
- [Result] Murthy V, Maitre P, Bakshi G, Pal M, Singh M, Sharma R, Gudipudi D, Pujari L, Pandey H, Bandekar B, Joseph D, Krishnatry R, Phurailatpam R, Kannan S, Arora A, Misra A, Joshi A, Noronha V, Prabhash K, Menon S, Prakash G. Bladder Adjuvant Radiation Therapy (BART): Acute and Late Toxicity From a Phase III Multicenter Randomized Controlled Trial. Int J Radiat Oncol Biol Phys. 2025 Mar 1;121(3):728-736. doi: 10.1016/j.ijrobp.2024.09.040. Epub 2024 Sep 29. PMID 39353477